CLINICAL TRIAL: NCT01915771
Title: A Phase 1, Open-label, Crossover Study to Determine the Intra-subject Variability of the Pharmacokinetics of Single Oral CapsuleDose of 20 mg Lomitapide in Healthy Subjects
Brief Title: Study to Determine the Intra-subject Variability of Pharmacokinetics of Lomitapide in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AEGR-733-026; 2013-002692-17 (EudraCT Number)
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Intra-subject Variability of Pharmacokinetics
MeSH Terms: interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lomitapide (Experimental): It will comprise of 2 single oral doses with at least a 14-day washout between doses.
  Interventions: Drug: lomitapide

INTERVENTIONS:
Drug: lomitapide — 20 mg dose
  Other Names: Juxtapid

SUMMARY:
Objectives:

To evaluate the intra-subject variability of the pharmacokinetics (PK) of single oral capsule doses of 20 mg lomitapide.

DETAILED DESCRIPTION:
This study will be a single centre, open-label study. It will comprise of 2 single oral doses with at least a 14-day washout between doses. Following the first dose subjects will be discharged from the unit for the remainder of the washout period. Subjects will be re-admitted to the unit on Day -1 (Period 2) and following an overnight fast they will be administered the second dose on Day 1 (Period 2). Subjects will be discharged from the unit following the 168 h PK blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a non-smoking healthy male or female, aged between 18 and 40 years of age.
2. Subject has a BMI of 18.5 - 25 kg/m2.
3. Subject has total body weight between > 50 kg to ≤ 100 kg.
4. Subjects must agree to use acceptable methods of contraception.
5. All females, regardless of childbearing potential, must have a negative serum beta human chorionic gonadotropin pregnancy test at Screening and on admission.
6. In good health, determined by no clinically significant or relevant abnormalities identified by a detailed medical history & full physical examination.
7. No known history of hypersensitivity or previous intolerance to lomitapide.
8. Subjects must be capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form prior to undergoing any study-related procedures.

Exclusion Criteria:

1. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion.
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
3. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations.
4. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
5. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) such as a QTcF interval of >450 msec, a history of a prolonged QTc interval or Brugada syndrome.
6. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, allergic, dermatological, metabolic, neurological, psychiatric or other disease.
7. History or laboratory evidence of Gilbert's syndrome.
8. Positive results in any of the serology tests for Hepatitis B Surface Antigen (HbsAg), anti-Hepatitis core antibody (anti-HBc Ig G [and anti-HBc IgM if IgG is positive], Hepatitis C antibodies (anti-HCV), and HIV 1 and 2 antibodies, (anti-HIV 1/2).
9. Use of any drugs of abuse within 6 months prior to admission.
10. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates and methadone) or from the alcohol breath test at screening and on admission (Day -1).
11. History or clinical evidence of alcohol or drug abuse within one year prior to admission.
12. Mentally handicapped.
13. Participation in a drug trial within 90 days prior to first drug administration.
14. Use of any prescription medication within 2 weeks prior to admission (Day -1), with the exception of the oral contraceptive pill.
15. Use of any substance inducing or inhibiting CYP3A4 enzymes within 30 days prior to admission (Day -1).
16. Use of any over-the-counter (OTC) medication (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to admission (Day -1), unless deemed acceptable by the Investigator and Sponsor.
17. Use of alcohol-, grapefruit-, starfruit-, or caffeine-containing foods or beverages within 72 hours prior to admission and through Study Completion.
18. Donation of more than 500 mL of blood within 90 days prior to drug administration.
19. Receipt of blood products within 2 months prior to admission.
20. Poor peripheral venous access.
21. Use of any tobacco- or nicotine-containing products within 6 months prior to admission (Day -1).
22. Any acute or chronic condition, scheduled hospitalisation (inclusive of elective surgery during study), or scheduled travel prior to completion of all study procedures.
23. Any circumstances or conditions, which, in the opinion of the PI, may affect full participation in the trial or compliance with the protocol.
24. Legal incapacity or limited legal capacity at screening.
25. Subjects who are vegetarians, vegans or have any dietary restrictions conflicting with the study standardised menus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2013-08-23 (Actual); Study Completion 2013-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sumeray, MD, Study Chair — Aegerion Pharmaceuticals, Inc.; Ulrike Lorch, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology, Croydon, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Day 1
Arm/Group | Lomitapide
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Day 15
Arm/Group | Lomitapide
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lomitapide
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum observed concentration of lomitapide and its metabolites, M1 & M3.
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: Only 13 subjects who had evaluable PK data in both study periods were included in the PK analysis of lomitapide. One subject was excluded from PK analysis of M1 and M3 during Period 1 due to early termination. Another subject was excluded from PK analysis of M1 and M3 during Period 2 because the subject did not complete both Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PK of Lomitapide: PK of Lomitapide Following a Single Oral Capsule Dose of 20 mg Lomitapide During Periods 1 and 2 (PK Set)
- PK of M1: PK of M1 Following a Single Oral Capsule Dose of 20 mg Lomitapide During Periods 1 and 2 (PK Set)
- PK of M3: PK of M3 Following a Single Oral Capsule Dose of 20 mg Lomitapide During Periods 1 and 2 (PK Set)
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
ng/mL
  Period 1 | 0.961 (0.556) | 2.34 (0.593) | 23.6 (7.08)
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 1.02 (0.843) | 2.20 (0.664) | 22.8 (9.33)

2. Primary Outcome: Tmax
Description: Time to reach maximum plasma concentration
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
hr
  Period 1 | 4.0 [1.00 to 18.0] | 5.00 [3.00 to 10.0] | 3.00 [1.00 to 4.03]
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 5.00 [3.00 to 18.0] | 5.00 [2.00 to 6.00] | 3.00 [1.00 to 4.00]

3. Primary Outcome: AUC0-t
Description: Area under the concentration-time curve from hour 0 to the last measurable concentration of lomitapide and its metabolites, M1 & M3.
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
ng*hr/mL
  Period 1 | 40.2 (18.1) | 65.8 (22.7) | 319 (153)
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 44.0 (21.7) | 62.8 (23.3) | 319 (176)

4. Primary Outcome: AUC0-∞
Description: Area under the concentration-time curve extrapolated to infinity for lomitapide and its metabolites, M1 & M3.
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
ng*hr/mL
  Period 1 | 44.4 (19.9) | 68.3 (23.6) | 330 (158)
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 48.3 (23.4) | 65.3 (24.1) | 330 (181)

5. Primary Outcome: λz
Description: Elimination rate constant estimated from individual linear regression of the terminal part of the log concentration vs time curve
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
1/hr
  Period 1 | 0.0141 (0.00196) | 0.0200 (0.00754) | 0.0155 (0.00370)
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 0.0146 (0.00139) | 0.0189 (0.00410) | 0.0172 (0.00272)

6. Primary Outcome: t1/2
Description: Apparent terminal elimination half-life
Time Frame: Pre dose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PK of Lomitapide | PK of M1 | PK of M3
Number analyzed (Participants) | 13 | 14 | 14
hr
  Period 1 | 50.3 (7.56) | 38.3 (10.6) | 46.9 (10.4)
  Period 2: number analyzed (Participants) | 13 | 13 | 13
  Period 2 | 47.8 (4.35) | 38.0 (6.61) | 41.2 (6.90)

ADVERSE EVENTS:
Groups:
- Period 1: All 15 subjects who were enrolled in the study received at least one 20 mg dose of lomitapide and had assessments for the analysis of safety during Period 1.
- Period 2: Only 13 subjects who were enrolled in the study received 2 single daily doses of 20 mg lomitapide as planned (one dose in each of the two study periods). 2 subjects who only received one dose in Period 1 due to early withdrawal were not included in analysis of safety during Period 2.
Arm/Group | Period 1 | Period 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 4/15 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (N=15) | Period 2 (N=13)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Lymphdenopathy (Blood and lymphatic system disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in contract